CLINICAL TRIAL: NCT05921305
Title: Randomized Trial of Mini-dose Methotrexate Plus Standard-dose Steroid vs Steroids for the Initial Treatment of Acute Graft Versus Host Disease
Brief Title: Mini-dose MTX Plus Standard-dose Steroid for the Initial Treatment of Acute GVHD
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Xiao-Jun Huang, director, hematology department,Peking University People's Hospital, Peking University People's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GVHD-MTX-Randomized trial
Record Dates: First submitted 2023-06-19; First posted 2023-06-27 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Acute Graft Versus Host Disease
MeSH Terms: interventions — Adrenal Cortex Hormones

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MTX and corticosteroid (Experimental): Methylprednisolone 2 mg/kg/day was given for 3 days, and for responding patients, the dose of prednisone must be at least 0.25mg/kg/day prednisone (or 0.2mg/kg/day methylprednisolone). MTX (5mg/m^2/day) was given on days 1, 3, and 8, and repeated weekly until aGVHD was CR.
  Interventions: Drug: MTX
- Corticosteroid (Active Comparator): Methylprednisolone 2 mg/kg/day was given for 3 days, and for responding patients, the dose of prednisone must be at least 0.25mg/kg/day prednisone (or 0.2mg/kg/day methylprednisolone).
  Interventions: Drug: Corticosteroid

INTERVENTIONS:
Drug: MTX — MTX (5mg/m^2/day) was given on days 1, 3, and 8, and repeated weekly until aGVHD was CR
  Arms: MTX and corticosteroid
Drug: Corticosteroid — Corticosteroid Methylprednisolone 2 mg/kg/day was given for 3 days, and for responding patients, the dose of prednisone must be at least 0.25mg/kg/day prednisone (or 0.2mg/kg/day methylprednisolone).
  Arms: Corticosteroid

SUMMARY:
This trial is a randomized (1:1) phase III open label study of frontline mini-MTX plus methylprednisolone 2mg/kg/day compared to methylprednisolone 2mg/kg in allogeneic stem cell transplant recipients with grade 2-4 aGVHD.

DETAILED DESCRIPTION:
Allo-HSCT is an effective treatment of malignant hematopoietic diseases. However, aGVHD remains a major complication after allo-HSCT. Corticosteroid is the standard first-line therapy for aGVHD. However, the response rate of corticosteroid was approximate 50%, and the clinical outcomes of patients with corticosteroid refractory GVHD were poor. Thus far, no combination therapy had been prove to be superior to corticosteroid alone as initial therapy for aGVHD. The study hypothesis: MTX combined corticosteroid treatment could help to control aGVHD.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who are fully informed and sign informed consent by themselves or their guardians;
2. Patients receiving first allogeneic hematopoietic stem cell transplantation;
3. Patients with acute graft-versus-host disease of grade II-IV were diagnosed after transplantation;
4. KPS>60, Estimated survival >3 months;
5. No serious organ damage:

   1. ANC in peripheral blood is greater than 0.5×109/l
   2. Creatinine < 1.5mg/dl
   3. Cardiac ejection index > 55%

Exclusion Criteria:

1. Patients with severe brain, heart, kidney or liver dysfunction unrelated to graft-versus host disease;
2. Patients with uncontrollable active infection;
3. Patients with recurrence of primary malignant hematopathy;
4. Expected survival is less than 3 months
5. Patients who have histories of severe allergic reactions
6. Pregnant or lactating women
7. The researcher judges that there are other factors that are not suitable for participating
8. Patients who received donor lymphocyte infusion

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 218 (Estimated)
Dates: Start 2023-08-03 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) for aGVHD treatment after treatment | 14 days
  Overall response rate is defined as the proportion of patients demonstrating a complete response or partial response without requirement for additional systemic therapies for an earlier progression, mixed response or non-response

SECONDARY OUTCOMES:
Overall response rate (ORR) for aGVHD treatment at 28 days after treatment | 28 days
  Overall response rate is defined as the proportion of patients demonstrating a complete response or partial response without requirement for additional systemic therapies for an earlier progression, mixed response or non-response
Overall response rate (ORR) for aGVHD treatment at 42 days after treatment | 42 days
  Overall response rate is defined as the proportion of patients demonstrating a complete response or partial response without requirement for additional systemic therapies for an earlier progression, mixed response or non-response
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 42 days
  Data collection including questionnaires at individual and group visits and physician interviews at individual visits will be used to assess participants for treatment-related adverse events.
cGVHD | 1 years
  The cumulative incidence of chronic GVHD
Infection and poor graft function | 1 year
  The cumulative incidence of severe infection and poor graft function
Relapse | 1 year
  The cumulative incidence of relapse
Non-relapse mortality | 1 year
  The cumulative incidence of non-relapse mortality
Overall survival | 1 year
  The cumulative incidence of overall survival
Disease free survival | 1 year
  The cumulative incidence of disease free survival

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Peking University Institute of Hematology,, Beijing, Beijing Municipality
  - Nanfang Hospital, Nanfang Medical University, Guangzhou, Guangdong

IPD SHARING:
Plan to Share IPD: No